CLINICAL TRIAL: NCT00484861
Title: The Effect of Diet on Vascular Disease: A Study of African American and Caucasian Women
Brief Title: Effect of Diet on Vascular Disease in Pre-Menopausal Women
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070163; 07-DK-0163
Record Dates: First submitted 2007-06-08; First posted 2007-06-11 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2017-02-14

CONDITIONS: Cardiovascular Diseases; Vascular Disease; Inflammation; Insulin; Triglycerides
Keywords: Women; Healthy Volunteers; Triglyceride; Healthy Volunteer; HV
MeSH Terms: conditions — Cardiovascular Diseases; Vascular Diseases; Inflammation; Insulin Resistance

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
African Americans have a higher prevalence of vascular disease than Caucasians. Vascular disease can lead to heart attacks, strokes and even amputations. Insulin, a hormone which is secreted by the pancreas, affects not only glucose and fat metabolism but also vascular disease. Impairment of insulin s ability to remove glucose from the circulation is known as insulin resistance. To overcome insulin resistance the pancreas secretes extra insulin. These high levels of insulin affect circulating triglyceride levels by both promoting production of triglyceride by the liver and interfering with clearance of triglyceride from the circulation. Triglyceride in turn contributes to the development of vascular disease by causing both inflammation and hypercoagulability.

Surprisingly African Americans are more insulin resistant and have a higher rate of vascular disease than Caucasians but have lower triglyceride levels. Because of the high rate of vascular diseases in African Americans, our aim is to determine if the adverse effects of triglyceride occur at a lower level in African Americans than Caucasians. To achieve this goal we will determine if there are differences in the effect of a meal on triglyceride levels and vascular function in a representative cohort of African American and Caucasian women.

For this study we will enroll 96 women (48 African American and 48 Caucasian women). We are recruiting women because ethnic differences in triglyceride are even greater in women than men. We are enrolling women between the ages of 18 and 65 years. The study will involve several outpatient visits to the NIH Clinical Center. The first visit will be a screening to determine eligibility. At the second visit a test to measure insulin resistance will be performed. This test is called a frequently sampled intravenous glucose tolerance test. The third visit will be for the test meal. Before and at 2, 4 and 6 hours after the meal, blood will be drawn and vascular function measured. Vascular function is determined by taking blood pressure and then measuring blood flow in the arm with ultrasound. It is possible that individual differences in diet could affect the results of the vascular study on the day of the test meal. Therefore for 7 days prior to the test meal, the NIH Clinical Center will provide to each participant all their meals in the form of either trays or meals in a box. These meals will be consistent with the typical American diet and be 33% fat, 15% protein and 52% carbohydrate. In designing these meals, the dietician will take into account individual food preferences.

This study is being performed in collaboration with the Harvard School of Public Health, the University of Texas Southwestern Medical Center and Indiana University. Therefore some blood drawn during Visits 2 and 3 will be sent coded, without personal identifiers, to each institution for analyses.

...

DETAILED DESCRIPTION:
African Americans have a higher prevalence of vascular disease than Caucasians. Vascular disease can lead to heart attacks, strokes and even amputations. Insulin, a hormone which is secreted by the pancreas, affects not only glucose and fat metabolism but also vascular disease. Impairment of insulin s ability to remove glucose from the circulation is known as insulin resistance. To overcome insulin resistance the pancreas secretes extra insulin. These high levels of insulin affect circulating triglyceride levels by both promoting production of triglyceride by the liver and interfering with clearance of triglyceride from the circulation. Triglyceride in turn contributes to the development of vascular disease by causing both inflammation and hypercoagulability.

Surprisingly African Americans are more insulin resistant and have a higher rate of vascular disease than Caucasians but have lower triglyceride levels. Because of the high rate of vascular diseases in African Americans, our aim is to determine if the adverse effects of triglyceride occur at a lower level in African Americans than Caucasians. To achieve this goal we will determine if there are differences in the effect of a meal on triglyceride levels and vascular function in a representative cohort of African American and Caucasian women.

For this study we will enroll 96 women (48 African American and 48 Caucasian women). We are recruiting women because ethnic differences in triglyceride are even greater in women than men. We are enrolling women between the ages of 18 and 65 years. The study will involve several outpatient visits to the NIH Clinical Center. The first visit will be a screening to determine eligibility. At the second visit a test to measure insulin resistance will be performed. This test is called a frequently sampled intravenous glucose tolerance test. The third visit will be for the test meal. Before and at 2, 4 and 6 hours after the meal, blood will be drawn and vascular function measured. Vascular function is determined by taking blood pressure and then measuring blood flow in the arm with ultrasound. It is possible that individual differences in diet could affect the results of the vascular study on the day of the test meal. Therefore for 7 days prior to the test meal, the NIH Clinical Center will provide to each participant all their meals in the form of either trays or meals in a box. These meals will be consistent with the typical American diet and be 33% fat, 15% protein and 52% carbohydrate. In designing these meals, the dietician will take into account individual food preferences.

This study is being performed in collaboration with the Harvard School of Public Health, the University of Texas Southwestern Medical Center and Indiana University. Therefore some blood drawn during Visits 2 and 3 will be sent coded, without personal identifiers, to each institution for analyses.

ELIGIBILITY:
* INCLUSION CRITERIA:

African American Women: Individuals will be considered to be African American if they self-identify as African American and were born in the United States. Further they must describe both parents as being African American.

Caucasian Women: Individuals will be considered to be Caucasian if they self-identify as Caucasian.

Healthy Volunteers: The potential enrollee must self identify as a normal volunteer and have this confirmed by having at the screening visit a normal complete blood count, glucose, BUN creatinine, liver and thyroid panel.

Age between 18 and 65 years: This age range is chosen because TG levels across the lifespan from early adulthood through to postmenopausal status. Weare using 65 years of age as a conventional upper limit. In addition, 65 years of age has been used as an age category cut-off by National Health and Nutrition Examination Surveys. Our goal is to detect ethnic differences in the pathways that allow vascular disease to develop. Enrolling women between the ages of 18 and 65 years, maximizes our ability to detect differences in mechanism of action that are truly secondary to ethnicity.

Weight less than 136 kg (300 lbs): This weight restriction is necessitated by the limitations of the DXA scanner. The DXA platform cannot accommodate subjects who weigh more than 136 kg.

BMI between 20 and 45 kg/m2: Women in both ethnic groups will be recruited across BMI nonobese and obese categories. Therefore we will enroll approximately equal numbers of women from each ethnic group in both BMI categories BMI between 20 and 30 kg/m(2) and BMI between 30 and 45 kg/m(2).

EXCLUSION CRITERIA:

Refusal to agree to use barrier contraception: The DXA scan and CT scan should not be performed if the participant is pregnant. In addition, TG levels are directly affected by pregnancy. Even though we will perform pregnancy tests within 7 days of each visit, we also require that the subject agree to abstinence or barrier contraception throughout the study.

Medications which affect parameters under investigation: Examples include corticosteroids, oral contraceptives, hypoglycemic (oral or injection), hypolipidemic, antihypertensive and antipsychotic agents. Oral contraceptives, in particular, are exclusion criteria because the estrogen component of oral contraceptives increase TG levels and would therefore obscure the effect of the test meal on TG levels.

Medical Conditions which affect parameters under investigation: Examples include diabetes, thyroid disease, liver disease, pancreatitis, nephrotic syndrome.

Hispanics: The relationship between TG and insulin resistance in Hispanic White women is midway between African American and Caucasian women. Therefore in this initial study to be able to determine the maximum ethnic difference in the relationship between TG and insulin resistance, we will enroll in this protocol study women who self-identify as African American and Caucasian and not enroll women who self-identify as Hispanic.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2007-06-07; Study Completion 2017-02-14

PRIMARY OUTCOMES:
Change in endothelial function after a meal.

SECONDARY OUTCOMES:
Ability of the presence or absence of insulin resistance to predict change in endothelial function after a meal.

CONTACTS AND LOCATIONS:
Overall Officials: Anne E Sumner, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ferdinand KC. Coronary artery disease in minority racial and ethnic groups in the United States. Am J Cardiol. 2006 Jan 16;97(2A):12A-19A. doi: 10.1016/j.amjcard.2005.11.011. Epub 2005 Dec 1. PMID 16442932
- [Background] Schwartz EA, Reaven PD. Molecular and signaling mechanisms of atherosclerosis in insulin resistance. Endocrinol Metab Clin North Am. 2006 Sep;35(3):525-49, viii. doi: 10.1016/j.ecl.2006.06.005. PMID 16959584
- [Background] Kissebah AH, Alfarsi S, Adams PW, Wynn V. Role of insulin resistance in adipose tissue and liver in the pathogenesis of endogenous hypertriglyceridaemia in man. Diabetologia. 1976 Dec;12(6):563-71. doi: 10.1007/BF01220632. PMID 187517
- [Derived] Wang L, Sacks FM, Furtado JD, Ricks M, Courville AB, Sumner AE. Racial differences between African-American and white women in insulin resistance and visceral adiposity are associated with differences in apoCIII containing apoAI and apoB lipoproteins. Nutr Metab (Lond). 2014 Dec 17;11(1):56. doi: 10.1186/1743-7075-11-56. eCollection 2014. PMID 25553059
- [Derived] Sumner AE, Thoreson CK, O'Connor MY, Ricks M, Chung ST, Tulloch-Reid MK, Lozier JN, Sacks DB. Detection of abnormal glucose tolerance in Africans is improved by combining A1C with fasting glucose: the Africans in America Study. Diabetes Care. 2015 Feb;38(2):213-9. doi: 10.2337/dc14-1179. Epub 2014 Oct 22. PMID 25338926
- [Derived] Sumner AE, Furtado JD, Courville AB, Ricks M, Younger-Coleman N, Tulloch-Reid MK, Sacks FM. ApoC-III and visceral adipose tissue contribute to paradoxically normal triglyceride levels in insulin-resistant African-American women. Nutr Metab (Lond). 2013 Dec 23;10(1):73. doi: 10.1186/1743-7075-10-73. PMID 24365086